CLINICAL TRIAL: NCT04786834
Title: Proficiency Based Progression Training Versus the Halsted's Model for a Robotic Vesico-urethral Anastomosis on an Avian Tissue Model: a Prospective, Randomized, Multicenter and Blinded Clinical Trial: the PROVESA Trial
Brief Title: PBP Versus Halsted's Model: the PROVESA Trial
Acronym: PROVESA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stefano Puliatti (Other)
Responsible Party: Sponsor-Investigator, Stefano Puliatti, Deputy Medical Director, Orsi Academy
Organization: Orsi Academy (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: PROVESA
Record Dates: First submitted 2021-01-09; First posted 2021-03-08 (Actual); Last update posted 2021-03-08 (Actual); Status verified 2021-03

CONDITIONS: Educational Problems
Keywords: surgery; robotics; training; vesico-urethral anastomosis; Proficiency Based Progression; Basic skills training

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Traditional training group (Active Comparator): Trainees in the Traditional trained group will be trained according to the traditional approach of 'See one, do one, teach one' principle. Trainees will have an e-learning didactic component (specifically on the anatomy & physiology of the procedure, clinical aspects of the procedure, published evidence etc) which they must complete before training by a procedure expert. On completion of the e-learning module they will complete a summative assessment of their knowledge. They will then be shown how and then trained to suture and tie knots using the robot. The VUA will be demonstrated initially by an expert and who will then proctor the trainees in the same technique for repeated training trials., i.e., repeated practice for a period of time matched to the PBP group.
  Interventions: Procedure: Vesico urethral anastomosis on chicken model
- Proficiency based progression (PBP) training group: a new training methodology (Experimental): Participants in the PBP trained group will follow the exact same e-learning didactic course as the Traditional trained group but the PBP group will be required to pass a test of procedure knowledge before continuing to the surgical training. Their knowledge will be assessed in a formative and summative fashion. After their initial VUA assessment, procedure-specific and validated procedure metrics will be used to teach the students the steps of the procedure, as well as the correct (and incorrect) way to perform the procedure. The metrics will be used to give them performance feedback with specific advice on how they might improve their performance, i.e., deliberate practice.
  Interventions: Procedure: Vesico urethral anastomosis on chicken model

INTERVENTIONS:
Procedure: Vesico urethral anastomosis on chicken model — Performance of a vesico urethral anastomosis on a chicken model with Da Vinci robotic system

SUMMARY:
This randomized controlled trial aims to compare the effectiveness of Halsted's apprenticeship approach to training with the PBP approach for teaching the robotic suturing of a VUA on a chicken model.

DETAILED DESCRIPTION:
In a prospective, randomized and blinded study robotic naïve (urology (n = 12), surgery (n = 12) and gynecology (n = 12)) residents (n = 36) from the KU Leuven and University of Gent residency training programs will be randomized (in equal discipline numbers) to Traditional Halstedian apprenticeship type training or proficiency based progression (PBP) training to learn to perform a vesico-urethral anastomosis (VUA) on a chicken model. Both groups will receive the same e-learning (on how to perform the VUA on the chicken model) and skills laboratory robotic training curriculum. The PBP trained group will however be required to demonstrate quantitively defined proficiency benchmarks for training progression (i.e., from e-learning to the skills lab). The PBP group will also have a defined benchmark to demonstrate before training is deemed completed. The Traditional trained group will train in the same skills laboratory for a case-matched period of time as the PBP group, with the same level of supervising faculty proctors and using the same training resources but with no proficiency benchmarks or metric-based feedback. Both groups will be required to perform a VUA on the chicken model before skills training proper and at the end of training. Investigators will be trained in pairs to assess VUA performance from a pre-defined set of explicitly defined binary metric events reliably (inter-rater reliability > 0.8). They will also be blinded as to the identity of the trainee performing the procedure, how they were trained (i.e., group) and procedure order.

H1 It is hypothesized that implementation of PBP training in teaching the robotic suturing of VUA leads to better surgical training outcomes (i.e., lower number of performance errors) when compared to Halsted's method.

ELIGIBILITY:
Inclusion Criteria:

* recently accepted, first or second year residents gynecology and obstetrics (n=12), urology (n=12) and general surgery (n=12). Novice in robotic surgery.

Exclusion Criteria:

* Any robotic experience

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2020-07-27 (Actual); Primary Completion 2020-08-15 (Actual); Study Completion 2020-08-15 (Actual)

PRIMARY OUTCOMES:
Surgical proficiency level determined by objectively assessed, validated, binary performance operative metrics. Comparison between PBP training versus traditional training for a robotic suturing and knot tying task. | 1 year
  The aim of this paper is to report the main outcomes of the PROVESA trial without emphasizing the interspecialty differences. The investigators will however emphasize its methodology, the fact that is well controlled and multicentric. Differences in proficiency level, assessed by binary performance metrics based assessment of a robotic suturing and knot tying task, will be reported.

SECONDARY OUTCOMES:
Cross-specialty differences in surgical proficiency levels, assessed by objectively assessed, validated, binary performance operative metrics, for a robotic suturing and knot tying task. | 1 year
  Surgical skill is often thought to be associated to surgical discipline. The aim of this study is to compare the objectively assessed training outcomes of different surgical disciplines (Surgery, Gynecology/obstetrics and Urology) performing the robotic suturing of a vesico-urethral anastomosis (VUA) on a chicken model. Participants were trained according to a traditional versus a proficiency based progression methodology and were assessed by the use of validated, binary performance operative metrics.
Difference in interrater reliability for metrics-based scoring determined by objectively assessed, validated, binary performance operative metrics versus GEARS-based scoring of a robotic suturing and knot tying task. | 2 years
  Nowadays, different methods are used to assess surgical performance. One of the most commonly used methods is the GEARS (Global Evaluative Assessment of Robotic Skills). This is, however, a qualitative scoring method which uses a Likert scale for scoring and which might be prone to poor interrater reliability and subjectiveness.
  The aim of this paper will be to report the interrater reliability of both scoring methods and the correlation between each other. Hypothesis is that interrater reliability will be superior for performance metrics. The investigators will try to answer the question which is the best tool to assess surgical performance.
Trainee's satisfaction as assessed by questionnaire with Likert scale. Does it influence outcome of surgical training? Comparison between proficiency based progression training versus traditional training for a robotic suturing and knot tying task. | 2 years
  Satisfaction of a surgical trainee is often thought to be key for training quality and a predictor of good outcome of surgical training. At the end of the PROVESA, all participants were asked to complete an online questionnaire where their satisfaction with the adopted training method was asked for using a Likert scale.
  Hypothesis is that trainee's satisfaction does NOT correlate with training outcome and that satisfaction is NOT a good determinator of training quality.
Correlation between live and video-based scoring of surgical performance | 2 years
  Surgical performance is often assessed live during surgery. However, one might miss specific details of performance. A possible answer to this query lies in video-based scoring of a surgical task. However, does video-based scoring reflects the same surgical quality? Moreover, one could question the ethical aspect of non-live scoring of surgical performance.
  In the PROVESA trial, all surgical tasks were scored live and video-based afterwards. The correlation in metrics-based performance scores between live and video-based assessment will be investigated.
  Hypothesis is that there will be no differences. The investigators will try to answer the question which scoring method will give the trainee the highest chance of reaching proficiency?
Reporting the outcome of the e-learning scores from an online proficiency questionnaire on an online learning platform. Comparison between proficiency based progression training versus traditional training for a robotic suturing and knot tying task. | 2 years
  During the PROVESA trial, all participants had to do an online assessment. This was done on an online learning platform using a questionnaire. A proficiency benchmark was set based on the mean score of experts on the same questionnaire.
  The PBP group needed to do this after doing an online curriculum during which the operative metrics were explained. In order to move forward to the clinical training in the lab, they had to show proficiency on the test by reaching a pre-defined benchmark.
  The Control group needed to do the online assessment after their day of training and after performing the final VUA. The investigators noted a significant correlation between the score on the online assessment and the number of metrics-based performance errors. The lower the score on the online test, the more performance errors they made.
  The aim of this paper will be to stipulate the importance of e-learning and online scoring and its correlation with surgical performance.

CONTACTS AND LOCATIONS:
Overall Officials: Ruben De Groote, MD, Principal Investigator — Orsi Academy
Locations (1):
- Orsi Academy, Melle, Oost-Vlaanderen, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Pellegrini CA. Surgical education in the United States: navigating the white waters. Ann Surg. 2006 Sep;244(3):335-42. doi: 10.1097/01.sla.0000234800.08200.6c. No abstract available. PMID 16926559
- [Result] Cuschieri A. Whither minimal access surgery: tribulations and expectations. Am J Surg. 1995 Jan;169(1):9-19. doi: 10.1016/s0002-9610(99)80104-4. No abstract available. PMID 7818004
- [Result] Gallagher AG. Metric-based simulation training to proficiency in medical education:- what it is and how to do it. Ulster Med J. 2012 Sep;81(3):107-13. PMID 23620606
- [Result] Gallagher AG, Ritter EM, Champion H, Higgins G, Fried MP, Moses G, Smith CD, Satava RM. Virtual reality simulation for the operating room: proficiency-based training as a paradigm shift in surgical skills training. Ann Surg. 2005 Feb;241(2):364-72. doi: 10.1097/01.sla.0000151982.85062.80. PMID 15650649
- [Result] Breen D, O'Brien S, McCarthy N, Gallagher A, Walshe N. Effect of a proficiency-based progression simulation programme on clinical communication for the deteriorating patient: a randomised controlled trial. BMJ Open. 2019 Jul 9;9(7):e025992. doi: 10.1136/bmjopen-2018-025992. PMID 31289064
- [Result] Kallidaikurichi Srinivasan K, Gallagher A, O'Brien N, Sudir V, Barrett N, O'Connor R, Holt F, Lee P, O'Donnell B, Shorten G. Proficiency-based progression training: an 'end to end' model for decreasing error applied to achievement of effective epidural analgesia during labour: a randomised control study. BMJ Open. 2018 Oct 15;8(10):e020099. doi: 10.1136/bmjopen-2017-020099. PMID 30327396
- [Result] Angelo RL, Ryu RK, Pedowitz RA, Beach W, Burns J, Dodds J, Field L, Getelman M, Hobgood R, McIntyre L, Gallagher AG. A Proficiency-Based Progression Training Curriculum Coupled With a Model Simulator Results in the Acquisition of a Superior Arthroscopic Bankart Skill Set. Arthroscopy. 2015 Oct;31(10):1854-71. doi: 10.1016/j.arthro.2015.07.001. Epub 2015 Sep 2. PMID 26341047
- [Result] Van Sickle KR, Ritter EM, Baghai M, Goldenberg AE, Huang IP, Gallagher AG, Smith CD. Prospective, randomized, double-blind trial of curriculum-based training for intracorporeal suturing and knot tying. J Am Coll Surg. 2008 Oct;207(4):560-8. doi: 10.1016/j.jamcollsurg.2008.05.007. Epub 2008 Jul 14. PMID 18926460
- [Result] Ahlberg G, Enochsson L, Gallagher AG, Hedman L, Hogman C, McClusky DA 3rd, Ramel S, Smith CD, Arvidsson D. Proficiency-based virtual reality training significantly reduces the error rate for residents during their first 10 laparoscopic cholecystectomies. Am J Surg. 2007 Jun;193(6):797-804. doi: 10.1016/j.amjsurg.2006.06.050. PMID 17512301
- [Result] Seymour NE, Gallagher AG, Roman SA, O'Brien MK, Bansal VK, Andersen DK, Satava RM. Virtual reality training improves operating room performance: results of a randomized, double-blinded study. Ann Surg. 2002 Oct;236(4):458-63; discussion 463-4. doi: 10.1097/00000658-200210000-00008. PMID 12368674
- [Result] Vanlander AE, Mazzone E, Collins JW, Mottrie AM, Rogiers XM, van der Poel HG, Van Herzeele I, Satava RM, Gallagher AG. Orsi Consensus Meeting on European Robotic Training (OCERT): Results from the First Multispecialty Consensus Meeting on Training in Robot-assisted Surgery. Eur Urol. 2020 Nov;78(5):713-716. doi: 10.1016/j.eururo.2020.02.003. Epub 2020 Feb 21. PMID 32089358
- [Result] Cacciamani G, De Marco V, Siracusano S, De Marchi D, Bizzotto L, Cerruto MA, Motton G, Porcaro AB, Artibani W. A new training model for robot-assisted urethrovesical anastomosis and posterior muscle-fascial reconstruction: the Verona training technique. J Robot Surg. 2017 Jun;11(2):123-128. doi: 10.1007/s11701-016-0626-4. Epub 2016 Jul 20. PMID 27440232
- [Result] Santos DRD, Calvo FC, Feijo DH, Araujo NP, Teixeira RKC, Yasojima EY. New training model using chickens intestine for pediatric intestinal anastomosis. Acta Cir Bras. 2019 Sep 16;34(7):e201900709. doi: 10.1590/s0102-865020190070000009. PMID 31531529
- [Result] Sotelo RJ, Astigueta JC, Carmona OJ, De Andrade RJ, Moreira OE. Chicken gizzard: a new training model for laparoscopic urethrovesical anastomosis. Actas Urol Esp. 2009 Nov;33(10):1083-7. doi: 10.1016/s0210-4806(09)73185-7. English, Spanish. PMID 20096178
- [Result] Ericsson KA. Towards a science of the acquisition of expert performance in sports: Clarifying the differences between deliberate practice and other types of practice. J Sports Sci. 2020 Jan;38(2):159-176. doi: 10.1080/02640414.2019.1688618. Epub 2019 Nov 12. PMID 31718526
- [Result] Goh AC, Goldfarb DW, Sander JC, Miles BJ, Dunkin BJ. Global evaluative assessment of robotic skills: validation of a clinical assessment tool to measure robotic surgical skills. J Urol. 2012 Jan;187(1):247-52. doi: 10.1016/j.juro.2011.09.032. Epub 2011 Nov 17. PMID 22099993
- [Result] Gallagher AG, Ritter EM, Satava RM. Fundamental principles of validation, and reliability: rigorous science for the assessment of surgical education and training. Surg Endosc. 2003 Oct;17(10):1525-9. doi: 10.1007/s00464-003-0035-4. Epub 2003 Sep 19. No abstract available. PMID 14502403

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-07-27): https://cdn.clinicaltrials.gov/large-docs/34/NCT04786834/Prot_SAP_000.pdf
  • Informed Consent Form (2020-07-27): https://cdn.clinicaltrials.gov/large-docs/34/NCT04786834/ICF_001.pdf